CLINICAL TRIAL: NCT01090791
Title: Assessment of the FLOTRAC/VIGILEO Third Generation Software to Predict Fluid Responsiveness in Critically Ill Patient With Acute Circulatory Failure
Brief Title: FLOTRAC/VIGILEO in Acute Circulatory Failure
Acronym: FLOVAC
Status: Terminated | Type: Observational
Why Stopped: Major change in protocol anticipated
Sponsor: Hôpital Européen Marseille (Other)
Responsible Party: Principal Investigator, Jerome Allardet-Servent, MD, MD, MSc, Hôpital Européen Marseille
Other Study IDs: 2009-A007419-48
Record Dates: First submitted 2010-03-22; First posted 2010-03-23 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Critically Ill; Acute Circulatory Failure; Fluid Loading
Keywords: critically ill patient
MeSH Terms: conditions — Critical Illness; Shock | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Flotrac/Vigileo third generation software — Measurement of stroke volume according to the arterial pressure waveform
Device: Transthoracic echocardiography — Measurement of stroke volume according to the aortic time-velocity integral

SUMMARY:
Acute circulatory failure may be related to hypovolemia. Fluid loading increases stroke volume in approximatively half of challenges. Determining fluid responsiveness prevents unnecessary fluid loading. Passive leg raising (PLR) provides a transient increase of 300 ml in venous return for a short time. The measurement of stroke volume (SV) before and after a PLR test allows physician to detect fluid responsiveness, when stroke volume increases is higher than 15 %. Beside thermodilution, the use of non invasive device to measure stroke volume becomes largely employed. Arterial Pressure based Cardiac Output (APCO), provided by the Flotrac/Vigileo system, does not required specific materials nor repeated calibration. The third generation software is believed to be more accurate and more precise for SV measurement. The aim of this study is to test the performance of the Flotrac/Vigileo device in a situation of rapid venous return changes induced by PLR and then by fluid loading. Patients will be classify posteriorly in responders and non responders, according to the magnitude of the fluid loading-induced SV changes measured by transthoracic echocardiography.

ELIGIBILITY:
Inclusion Criteria:

* Systolic arterial pressure < 90 mmHg or Mean arterial pressure < 60 mmHg
* Heart rate > 100 bpm
* Norepinephrine infusion
* Urine output < 0.5 ml/kg/h during at least two consecutive hours
* skin mottling
* Capillary refill time > 3 sec

Exclusion Criteria:

* Acute cor pulmonale
* Ongoing renal replacement therapy
* Lack of echogenicity during transthoracic echocardiography

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients with acute circulatory failure, as defined by two or more of the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2011-05; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Stroke volume measurement between Flotrac/Vigileo device and transthoracic echocardiography | 30 min
  Bland-Altman analysis of the whole SV measurements

SECONDARY OUTCOMES:
SV cut-off with Flotrac/Vigileo and with TEE to predict fluid responsiveness | 30 min
  ROC curve
SVV cut-off with Flotrac/Vigileo to predict fluid responsiveness | 30 min
  ROC curve

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme Allardet-Servent, MD,MSc, Principal Investigator — Fondation Hôpital Ambroise Paré
Locations (2):
- France (2):
  - Hopital Paul Desbief, Marseille
  - Hopital Ambroise Paré, Marseille